CLINICAL TRIAL: NCT02738489
Title: An Open-Label, Single Center, Nonrandomized, Dose-Escalation Phase 1 Study to Evaluate Safety and Tolerability of SHR-1210 in Subjects With Advanced Melanoma
Brief Title: A Study to Evaluate the Safety and Tolerability of Using the SHR-1210 in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-102
Record Dates: First submitted 2016-04-10; First posted 2016-04-14 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Advanced Melanoma
Keywords: PD-1/PD-L1 Advanced Melanoma Immunotherapy
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Injection SHR-1210 60mg Cohort (Experimental)
  Interventions: Biological: SHR-1210
- Injection SHR-1210 200mg Cohort (Experimental)
  Interventions: Biological: SHR-1210
- Injection SHR-1210 400mg Cohort (Experimental)
  Interventions: Biological: SHR-1210

INTERVENTIONS:
Biological: SHR-1210 — A fully human monoclonal immunoglobulin (IgG4 subtype)

SUMMARY:
This is an open-label, single center, non-randomized, dose escalation phase I trial to evaluate safety and tolerability of SHR-1210 (camrelizumab) in patients with advanced melanoma with disease progression after standard treatment, unresectable lesions, or metastases. Between Apr 13, 2016, and Jan 8, 2020, 36 patients were enrolled from Beijing Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 years old, who agree to provide pathological tumor biopsy specimens during the screening period and after the end of treatment.
2. Patients with pathologically confirmed advanced melanoma who have failed standard treatments or without effective treatment methods (e.g., chemotherapy, targeted therapy and immunotherapy other than those targeting PD-1/PD-L1).
3. ECOG PS: 0-1.
4. Life expectancy ≥ 12 weeks.
5. With measurable and evaluable lesion(s) according to RECIST v1.1.

Exclusion Criteria:

1. Patients with active autoimmune diseases or a history of autoimmune diseases (including but not limited to the following: interstitial pneumonitis, uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism; adults with vitiligo or completely relieved childhood asthma can be enrolled if they do not require any intervention; patients with asthma requiring medical intervention with bronchodilators cannot be enrolled).
2. Patients who are currently using immunosuppressive agents, or systemic or absorbable local hormonal therapies for immunosuppression purposes (> 10 mg/day prednisone or equivalent) and still use the above drugs within 2 weeks prior to enrollment.
3. Patients who are known to be previously allergic to macromolecular protein preparations or any component of SHR-1210.
4. Patients with clinically symptomatic metastases to central nervous system (e.g., cerebral edema requiring hormonal intervention, or progression of brain metastasis). Patients who have received treatment for brain or meningeal metastasis can be included if they are clinically stable (MRI) for at least 2 months and have discontinued systemic hormonal therapy (> 10 mg/day prednisone or equivalent) for more than 2 weeks.
5. Patients who have previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy with an interval of less than 4 weeks from the completion of the treatment to the study medication (for patients who have previously received chemotherapy with nitrosourea or mitomycin, the interval from the end of chemotherapy to the study enrollment is less than 6 weeks); patients whose adverse events caused by previous treatments have not recovered to CTCAE Grade ≤ 1.
6. Patients with active infection or unexplained fever > 38.5 °C during screening or prior to the first dose (patients with tumor-induced fever may be enrolled as per the judgment of the investigator).
7. Patients with congenital or acquired immunodeficiency (such as HIV, HBV, or HCV).
8. Patients who have previously received other PD-1 antibody treatments or immunotherapies targeting PD-1/PD-L1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | From the time the participants signed the informed consent to 90 days after the final dose (Up to 3 years and 9 months)
  The safety assessment documented in this clinical study included any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an investigational product, which were monitored per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version [v] 4.03 2010).
Number of Participants Experiencing Severe AEs (SAEs) | From the time the participants signed the informed consent to 90 days after the final dose (Up to 3 years and 9 months)
  The safety assessment documented in this clinical study included any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an investigational product, which were monitored per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version [v] 4.03 2010).

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) For SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Area Under the Serum Concentration-time Curve to infinite time (AUC 0-inf) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Area Under the Serum Concentration-time Curve from dosing to the time of the last measured concentration (AUC 0-last) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Time to Maximum Concentration (Tmax) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Half-life (T½) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Clearance (Cl) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Volume of distribution (Vd) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Mean Residence Time (MRT) for SHR-1210 | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
C(ss, Max) of SHR-1210 after Multiple Dosing | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
C(ss, Min) of SHR-1210 after Multiple Dosing | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
Accumulation ratio based on Cmax (Rac, Cmax) of SHR-1210 after Multiple Dosing | PK blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
PD-1 receptor occupancy (RO) for SHR-1210 | PD blood samples are collected multiple times on Cycle 1 (each cycle is 28 days) Day1, Day 8, Day 15, Day 22, Cycle 2 Day 1, Since Cycle 2, every 3 cycle Day 1, and the day disease progression (Up to 3 years and 9 months).
  Receptor occupancy (RO) assays are designed to quantify the binding of therapeutics to their targets on the cell surface and are frequently used to generate pharmacodynamic (PD) biomarker data in nonclinical and clinical studies of biopharmaceuticals.
Number of Participants with Anti-drug Antibodies (ADAs) for SHR-1210 | Blood samples for ADAs analysis are collected on Cycle 1 (each cycle is 28 days) Day1 to the end of treatment (Up to 3 years and 9 months).
  ADAs: Immunogenicity was summarized by the number and percentage of participants who developed detectable treatment-emergent ADAs.
Objective Response Rate (ORR) | Up to 3 years and 9 months
  ORR was defined as the percentage of participants in the study whose best overall response was either complete response (CR) or partial response (PR) as assessed by investigators based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
Disease Control Rate (DCR) | Up to 3 years and 9 months
  DCR was defined as the percentage of participants in the study whose best overall response was either CR, PR or stable disease (SD) as assessed by investigators based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
Progression-free survival (PFS) | Up to 3 years and 9 months
  PFS was defined as the time from the date of first study dose to disease progression or death whichever occurs first. Participants without an event (no disease progression or death) were censored at the date of "last tumor assessment". Participants with no baseline or post-baseline tumor assessments were censored at Day 1. PFS was based on RECIST v 1.1 and the results of Investigator evaluations. Median PFS was calculated by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Yiding Xing, Doctor, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (1):
- Cancer Hospital Affiliated to Beijing University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou L, Wu X, Chi Z, Si L, Sheng X, Kong Y, Mao L, Lian B, Tang B, Yan X, Wang X, Bai X, Li S, Wei X, Li J, Yang Q, Guo J, Cui C. Safety, activity, and pharmacokinetics of camrelizumab in advanced Asian melanoma patients: a phase I study. BMC Cancer. 2022 May 20;22(1):565. doi: 10.1186/s12885-022-09663-5. PMID 35596181